CLINICAL TRIAL: NCT03421782
Title: Nonpharmacologic Interventions for Fatigue in Patients With Cancer
Brief Title: Fatigue Interventions in Cancer (Exercise Intervention)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI105691; NCI-2017-02424 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Sedentary Lifestyle; Stage III Prostate Cancer AJCC v7; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Sedentary Behavior; Prostatic Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise - Arm I (Experimental): Patients undergo POWER exercise intervention consisting of supervised exercise training sessions over 50 minutes every 7 days for a total of 12 sessions and 150 minutes of moderate-intensity exercise weekly for 12 weeks.
  Interventions: Behavioral: Exercise Intervention
- Exercise plus PROSPECT Cognitive Behavior Therapy (CBT) (Experimental): Patients undergo POWER exercise intervention consisting of supervised exercise training sessions over 50 minutes every 7 days for a total of 12 sessions and 150 minutes of moderate-intensity exercise weekly for 12 weeks. Patients also undergo PROSPECT internet-based CBT intervention over 12 weeks.
  Interventions: Behavioral: Cognitive Behavior Therapy; Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Undergo PROSPECT internet-based CBT
  Other Names: CBT; cognitive therapy; CT
  Arms: Exercise plus PROSPECT Cognitive Behavior Therapy (CBT)
Behavioral: Exercise Intervention — Undergo POWER exercise intervention

SUMMARY:
This randomized pilot phase II trial studies how well exercise intervention with or without internet-based cognitive behavior therapy works in reducing fatigue in participants with prostate cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Exercise intervention and internet-based cognitive behavior therapy may help to improve feelings of tiredness in participants with prostate cancer.

The study originally included both prostate cancer and breast cancer participants, but due to low accrual of breast cancer participants, the breast cancer cohort was closed and the study continued with prostate cancer participants only.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the change in fatigue from baseline to week 12 in all patients with prostate cancer, as assessed with the PROMIS Fatigue questionnaire, with 12 weeks of POWER exercise program.

SECONDARY OBJECTIVES:

I. To evaluate the change in fatigue from baseline to week 12 in patients with prostate cancer who completed both baseline and 12 week assessments, as assessed with the PROMIS Fatigue questionnaire, with 12 weeks of the POWER exercise program.

II. To evaluate the change in cardiorespiratory fitness from baseline to Week 12, as assessed with the graded exercise test, with 12 weeks of the POWER exercise program.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo POWER exercise intervention consisting of supervised exercise training sessions over 50 minutes every 7 days for a total of 12 sessions and 150 minutes of moderate-intensity exercise weekly for 12 weeks.

ARM II: Patients undergo POWER exercise intervention consisting of supervised exercise training sessions over 50 minutes every 7 days for a total of 12 sessions and 150 minutes of moderate-intensity exercise weekly for 12 weeks. Patients also undergo PROSPECT internet-based cognitive behavior therapy (CBT) intervention over 12 weeks.

After completion of study, patients are followed up every 6-12 months for 2 years.

Because of challenges with the PROSPECT intervention, including multiple periods of time during which the intervention was not available and loss of data about use of the intervention by participants because of a computer virus, it appears that the majority of patients randomized to that arm of the study did not actually use the intervention. Therefore evaluable participants will be combined and analyzed as a single cohort.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with advanced prostate cancer
* Currently treated with hormone therapy-based regimen, including selective estrogen receptor modulators (SERMs), aromatase inhibitors, selective estrogen receptor down regulators (SERDs), CYP17A1 inhibitors, gonadotrophin releasing hormone (GnRH) agonists/antagonists, and antiandrogens; concurrent anti-HER2 therapy and other targeted therapy (e.g., CDK4/6 inhibitor, mTOR inhibitor) is permitted; must have started the current regimen at least 4 weeks prior to enrollment
* A response of at least 4 on a 10 point scale (with 0 = not tired at all and 10 = extremely tired) to the question ?how tired did you feel in the past week??
* Sedentary activity pattern (Average < 90 minutes per week of moderate-to-vigorous intensity sports activity based on patient self-report) within the past year
* Physically able to exercise and physician consent to start an exercise program
* Regular access to a computer with internet service
* Must be able to read and understand English
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Evidence of disease progression at the time of enrollment
* Treatment with cytotoxic chemotherapy within 3 months prior to enrollment
* Prior cognitive-behavioral therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Change in fatigue | Baseline up to 12 weeks post intervention (24 weeks)
  Change in fatigue from baseline to week 12 in all patients with prostate cancer, as assessed with the PROMIS Fatigue questionnaire, with 12 weeks of the POWER exercise program.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline up to 12 weeks post intervention (24 weeks)
  Change in fatigue from baseline to week 12 in patients with prostate cancer who completed both baseline and 12 week assessments, as assessed with the PROMIS Fatigue questionnaire, with 12 weeks of the POWER exercise program.
Change in activity level | Baseline up to 12 weeks post intervention (24 weeks)
  Evaluate the change in cardiorespiratory fitness from baseline to Week 12, as assessed with the graded exercise test, with 12 weeks of the POWER exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maughan, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States